CLINICAL TRIAL: NCT04823546
Title: Comparison of Effects of Activity Base Therapy vs Strength Training on Gait Performance in Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/20/2048 Anas Arshad
Record Dates: First submitted 2021-03-26; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Stroke
Keywords: Activity based therapy; Chronic stroke; Gait; strength training; exercises
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activity based therapy (Experimental): Activity based training was done in 2 phases. exercise involve
  1. Standing and reaching
  2. Sit-to-stand
  3. Stepping forward and backward Phase 2 Phase 2 started after 3 weeks. Phase 2 included the phase 1 exercise along with below exercise.
  (10) Walking on a treadmill;
  Interventions: Other: activity based therapy
- strength training (Active Comparator): Strength training for hip • flexor and extensors and abductors, knee extensors, and ankle dorsi flexors and plantar •flexors. Apart from using body weight, sandbag weights and Therabands of eight different resistances
  Interventions: Other: Strength Training

INTERVENTIONS:
Other: activity based therapy — Standing and reaching (2) Sit-to-stand (3) Stepping forward and backward onto blocks (4) Stepping sideways onto blocks (5) Forward step up onto blocks (6) Raising and lowering of heel (7) Standing with the base of support constrained with feet in parallel and tandem conditions Phase 2 started after 3 weeks. Phase 2 included the phase 1 exercise along with below exercise. (10) Walking on a treadmill; (11) Walking over various surfaces and obstacles;
  Arms: Activity based therapy
Other: Strength Training — Strength training included for hip • flexor and extensors and abductors, knee extensors, and ankle dorsi flexors and plantar •flexors. Apart from using body weight, sandbag weights and Therabands of eight different resistances
  Arms: strength training

SUMMARY:
Stroke is a leading cause of disability worldwide affecting both male and female especially in older people. Functional independence and locomotion are hampered in stroke, therefore, affecting their quality of life. Objective: To find the comparative effects of activity base therapy vs strength training on gait performance in chronic stroke patients.

DETAILED DESCRIPTION:
It was a randomized controlled trial, conducted in physical therapy department of Sir Ganga Ram Hospital. 20 chronic stroke patients were equally divided into two groups. In group-A patients were treated with activity base therapy and in group-B patients were treated with strength training. Patients were treated for a total of 6 weeks (12 sessions), 1 hour in a day, 3 times per week. Patients were assessed using Timed Up and Go (TUG) test and Fugl Meyer Examination-Lower Extremity (FME-LE). SPSS 25 was used toanalyze the dat

ELIGIBILITY:
Inclusion Criteria:

* Participants were at least 6 months post stroke.
* Ability to walk independent or with help of walking aids
* Ischemic stroke patients included in study.
* Mini mental state examination patients fully understand the commands

Exclusion Criteria:

* Presence of orthopaedic problems.

  * Neurological disorders.
  * Psychological problems.
  * Cognitive issues.
  * People with severe visual issues.
  * Participants with other medical complications foot ulcers, orthopaedic or other neurological impedance

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Time Up and Go Test (TUG) | 2 months
  Simple screening test that is a sensitive and specific measure of probability for falls among older adultsThe Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance.
  It uses the time that a person takes to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair, and sit down while turning 180 degrees.
Fugl meyer for lower limb | 2 months
  The fugal-meyer assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning in patient with post stroke hemiplegia.

CONTACTS AND LOCATIONS:
Overall Officials: Binash Afzal, PHD*, Principal Investigator — Riphah international university lahore campus
Locations (1):
- Binash afzal, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saleh MSM, Rehab NI, Aly SMA. Effect of aquatic versus land motor dual task training on balance and gait of patients with chronic stroke: A randomized controlled trial. NeuroRehabilitation. 2019;44(4):485-492. doi: 10.3233/NRE-182636. PMID 31256082
- [Background] Tisserand R, Armand S, Allali G, Schnider A, Baillieul S. Cognitive-motor dual-task interference modulates mediolateral dynamic stability during gait in post-stroke individuals. Hum Mov Sci. 2018 Apr;58:175-184. doi: 10.1016/j.humov.2018.01.012. Epub 2018 Mar 12. PMID 29448162
- [Background] Park HK, Lee HJ, Lee SJ, Lee WH. Land-based and aquatic trunk exercise program improve trunk control, balance and activities of daily living ability in stroke: a randomized clinical trial. Eur J Phys Rehabil Med. 2019 Dec;55(6):687-694. doi: 10.23736/S1973-9087.18.05369-8. Epub 2018 Oct 29. PMID 30370752
- [Background] Lund C, Dalgas U, Gronborg TK, Andersen H, Severinsen K, Riemenschneider M, Overgaard K. Balance and walking performance are improved after resistance and aerobic training in persons with chronic stroke. Disabil Rehabil. 2018 Oct;40(20):2408-2415. doi: 10.1080/09638288.2017.1336646. Epub 2017 Jun 9. PMID 28597708
- [Background] Lee HS, Park YJ, Park SW. The Effects of Virtual Reality Training on Function in Chronic Stroke Patients: A Systematic Review and Meta-Analysis. Biomed Res Int. 2019 Jun 18;2019:7595639. doi: 10.1155/2019/7595639. eCollection 2019. PMID 31317037
- [Background] Lamberti N, Straudi S, Malagoni AM, Argiro M, Felisatti M, Nardini E, Zambon C, Basaglia N, Manfredini F. Effects of low-intensity endurance and resistance training on mobility in chronic stroke survivors: a pilot randomized controlled study. Eur J Phys Rehabil Med. 2017 Apr;53(2):228-239. doi: 10.23736/S1973-9087.16.04322-7. Epub 2016 Sep 14. PMID 27626795
- [Background] Vahlberg B, Cederholm T, Lindmark B, Zetterberg L, Hellstrom K. Short-term and long-term effects of a progressive resistance and balance exercise program in individuals with chronic stroke: a randomized controlled trial. Disabil Rehabil. 2017 Aug;39(16):1615-1622. doi: 10.1080/09638288.2016.1206631. Epub 2016 Jul 14. PMID 27415645
- [Background] Wist S, Clivaz J, Sattelmayer M. Muscle strengthening for hemiparesis after stroke: A meta-analysis. Ann Phys Rehabil Med. 2016 Apr;59(2):114-24. doi: 10.1016/j.rehab.2016.02.001. Epub 2016 Mar 8. PMID 26969343
- [Background] Chan K, Phadke CP, Stremler D, Suter L, Pauley T, Ismail F, Boulias C. The effect of water-based exercises on balance in persons post-stroke: a randomized controlled trial. Top Stroke Rehabil. 2017 May;24(4):228-235. doi: 10.1080/10749357.2016.1251742. Epub 2016 Nov 3. PMID 27808012
- [Background] Geiger M, Supiot A, Zory R, Aegerter P, Pradon D, Roche N. The effect of transcranial direct current stimulation (tDCS) on locomotion and balance in patients with chronic stroke: study protocol for a randomised controlled trial. Trials. 2017 Oct 23;18(1):492. doi: 10.1186/s13063-017-2219-6. PMID 29061169